CLINICAL TRIAL: NCT00276848
Title: Fludarabine Versus Fludarabine Plus Cyclophosphamide in First Line Therapy of Younger Patients (Up to 65 Years) With Advanced Chronic Lymphocytic Leukemia (CLL)
Brief Title: Fludarabine With or Without Cyclophosphamide in Treating Patients With Advanced Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL4; EU-20538; GCLLSG-153; ISRCTN75653261; MEDAC-GCLLSG-CLL4; CDR0000455094 (Other: Clinical Data Repository)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fludarabine plus Cyclophosphamide (Active Comparator)
  Interventions: Drug: Fludarabine plus Cyclophosphamide
- Fludarabine (Active Comparator)
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: Fludarabine plus Cyclophosphamide — fludarabine at a dose of 25 mg/m2, administered intravenously daily over 30 minutes for 5 days, or fludarabine dosed at 30 mg/m2, administered intravenously daily over 30 minutes for 3 days, plus cyclophosphamide dosed at 250 mg/m2, administered intravenously daily over 30 minutes for 3 days, repeated every 28 days for a maximum of 6 courses
  Arms: Fludarabine plus Cyclophosphamide
Drug: Fludarabine — fludarabine at a dose of 25 mg/m2, administered intravenously daily over 30 minutes for 5 days, or fludarabine dosed at 30 mg/m2, administered intravenously daily over 30 minutes for 3 days, , repeated every 28 days for a maximum of 6 courses
  Arms: Fludarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving fludarabine together with cyclophosphamide is more effective than fludarabine alone in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying giving fludarabine together with cyclophosphamide to see how well it works compared to fludarabine alone in treating patients with advanced chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival, as well the overall survival and duration of remission in patients with previously untreated, advanced chronic lymphocytic leukemia treated with fludarabine with versus without cyclophosphamide.

Secondary

* Compare the incidence of side effects and quality of life of patients treated with these drugs.

OUTLINE: This is a multicenter, randomized study. Patients are randomized to 1 of 2 treatment arms

* Arm I: Patients receive fludarabine IV on days 1-5.
* Arm II: Patients receive fludarabine IV and cyclophosphamide IV on days 1-3. In both arms, treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 375 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of previously untreated chronic lymphocytic leukemia (CLL)

  * Binet stage C and stage B are acceptable if there is rapid disease progression, symptoms of enlarged lymph nodes and organs, or severe B-symptoms
  * Binet stage A is acceptable, if there are B-symptoms

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* No severe organ dysfunction
* No other previous or concurrent neoplasms, autoimmune hemolytic anemia, or thrombocytopenia

PRIOR CONCURRENT THERAPY:

* No prior or concurrent chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 1999-07; Primary Completion 2003-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 18 Month after end of treatment of the last patient
  date of randomization until progression of disease or death of any cause
Overall survival | 18 Month after end of treatment of the last patient
  Date of randomization until date of death
Duration of remission | 18 Month after end of treatment of the last patient
  Clinical response was defined according to the guidelines of the NCI-sponsored workshop

SECONDARY OUTCOMES:
Incidence of side effects | up to 28 days after the last dose of study medication
  Toxic effects of treatment were evaluated according to the Common Toxicity Criteria (CTC 1.0)
Quality of life | 18 Month after end of treatment of the last patient
  EORTC QUOL Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (134):
- Austria (2):
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
  - Hanuschkrankenhaus, Vienna
- Germany (132):
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Internistische Praxis - Arnstadt, Arnstadt
  - Specialist Practice for Oncology, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Kreiskrankenhaus, Bad Hersfeld
  - Caritas-Krankenhaus Bad Mergentheim, Bad Mergentheim
  - Humaine - Clinic, Bad Saarow
  - Internistische Praxis - Bad Salzuflen, Bad Salzuflen
  - Internistische Praxis - Bayreuth, Bayreuth
  - Internistische Gemeinschaftspraxis - Bergisch Gladbach, Bergisch Gladbach
  - Charite - Campus Charite Mitte, Berlin
  - Onkolog - Haematolog Schwerpunktpraxis, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Onkologische Gemeinschaftspraxis - Berlin, Berlin
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Evang. Waldkrankenhaus Spandau, Berlin
  - Internistische Praxis - Berlin, Berlin
  - Krankenhaus Bietigheim, Bietigheim
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Internistische Praxis - Chemnitz, Chemnitz
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Onkologische Schwerpunktpraxis, Cottbus
  - Onkologische Gemeinschaftspraxis - Dresden, Dresden
  - Krankenhaus Benrath, Düsseldorf
  - St. Georg Klinikum Eisenach GmbH, Eisenach
  - Hans - Susemihl - Krankenhaus, Emden
  - Internistische/Onkologische Praxis - Erfurt, Erfurt
  - Praxis DR. J. Weniger, Erfurt
  - Klinikum Erfurt, Erfurt
  - Praxis fuer Haematologie/Onkologie - Erfurt, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Onkologische Praxis - Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Internistische Gemeinschaftspraxis - Forchheim, Forchheim
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt
  - Gemeinschaftspraxis - Freiburg, Freiburg im Breisgau
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Internistische Praxis - Gerlingen, Gerlingen
  - Internistische Praxisgemeinschaft, Germering
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Klinik fuer Radioonkologie und Strahlentherapie, Göppingen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Praxis fuer Haematologie und Internistische Onkologie - Greifswald, Greifswald
  - Internistisch-Haematologische Gemeinschaftspraxis - Gustrow, Güstrow
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Internistische Praxis - Halle, Halle
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Schwerpunktpraxis Haematologie/Onkologie - Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - SLK - Kliniken Heilbronn GmbH - Klinikum am Gesundbrunnen, Heilbronn
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - Onkologische Schwerpunktpraxis, Hildesheim
  - Evang. Hospital, Holzminden
  - Universitaetsklinikum des Saarlandes, Homburg
  - Onkologische Gemeinschaftspraxis - Hoevelhof, Hövelhof
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Internistische Praxis - Ingolstadt, Ingolstadt
  - Internistische Gemeinschaftspraxis - Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Onkologische Gemeinschaftspraxis - Kaiserslautern, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius-Kliniken, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Klinikum Kempten Oberallgaeu, Kempten
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Klinikum Lippe - Lemgo, Lemgo
  - Internistische Praxis - Ludwigsburg, Ludwigsburg
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - III Medizinische Klinik Mannheim, Mannheim
  - Haematologische Praxis - Moenchengladbach, Mönchengladbach
  - Internistische Praxis - Muhr am See, Muhr am See
  - Klinikum der Universitaet Muenchen - Innenstadt Campus, Munich
  - Munich Oncologic Practice at Elisenhof, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Hamatologie/Onkologie Praxisgemeinschaft - Muenchen, München
  - University of Muenster, Münster
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Sudharz-Krankenhaus Nordhausen gGmbH, Nordhausen
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Paracelsus Karankenhaus Ruit, Ostfildern
  - Asklepios Klinik Pasewalk, Pasewalk
  - Vogtland - Klinikum Plauen GMBH, Plauen
  - Klinikum Ernst Von Bergmann, Postdam
  - Internistische Gemeinschaftspraxis - Potsdam, Potsdam
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Staedtische Klinikum-Kinderklinik, Rosenheim
  - Haematologische/Onkologische Schwerpunktpraxis - Rostock, Rostock
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbruecke
  - Caritasklinik St. Theresia, Saarbrücken
  - Klinikum Schwerin, Schwerin
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Internistische Gemeinschaftspraxis - Stuttgart, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Schwerpunktpraxis für Rheumatologie und Haematologie/Internistische Onkologie, Tübingen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Haematologisch-Onkologische Schwerpunktpraxis - Weilheim, Weilheim
  - Internistische Praxis - Wendlingen, Wendlingen
  - Gemeinschaftspraxis, Worms
  - Kliniken St. Antonius, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg
  - Internistische Praxis - Zittau, Zittau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichhorst BF, Fischer K, Fink AM, Elter T, Wendtner CM, Goede V, Bergmann M, Stilgenbauer S, Hopfinger G, Ritgen M, Bahlo J, Busch R, Hallek M; German CLL Study Group (GCLLSG). Limited clinical relevance of imaging techniques in the follow-up of patients with advanced chronic lymphocytic leukemia: results of a meta-analysis. Blood. 2011 Feb 10;117(6):1817-21. doi: 10.1182/blood-2010-04-282228. Epub 2010 Dec 7. PMID 21139079
- [Background] Cramer P, Bahlo J, Eichhorst B, Fischer K, Hallek M. Extramedullary manifestations of chronic lymphocytic leukaemia are not unusual. Leuk Res. 2014 Mar;38(3):284-5. doi: 10.1016/j.leukres.2013.11.015. Epub 2013 Dec 1. No abstract available. PMID 24412156
- [Background] Goede V, Cramer P, Busch R, Bergmann M, Stauch M, Hopfinger G, Stilgenbauer S, Dohner H, Westermann A, Wendtner CM, Eichhorst B, Hallek M; German CLL Study Group. Interactions between comorbidity and treatment of chronic lymphocytic leukemia: results of German Chronic Lymphocytic Leukemia Study Group trials. Haematologica. 2014 Jun;99(6):1095-100. doi: 10.3324/haematol.2013.096792. Epub 2014 Feb 28. PMID 24584349
- [Background] Jebaraj BMC, Tausch E, Landau DA, Bahlo J, Robrecht S, Taylor-Weiner AN, Bloehdorn J, Scheffold A, Mertens D, Bottcher S, Kneba M, Jager U, Zenz T, Wenger MK, Fingerle-Rowson G, Wendtner C, Fink AM, Wu CJ, Eichhorst B, Fischer K, Hallek M, Dohner H, Stilgenbauer S. Short telomeres are associated with inferior outcome, genomic complexity, and clonal evolution in chronic lymphocytic leukemia. Leukemia. 2019 Sep;33(9):2183-2194. doi: 10.1038/s41375-019-0446-4. Epub 2019 Mar 25. PMID 30911113
- [Background] Sachanas S, Pangalis GA, Fink AM, Bahlo J, Fischer K, Levidou G, Kyrtsonis MC, Bartzi V, Vassilakopoulos TP, Kalpadakis C, Koulieris E, Moschogiannis M, Yiakoumis X, Tsirkinidis P, Angelopoulou MK, Eichhorst B, Hallek M. Small Lymphocytic Lymphoma: Analysis of Two Cohorts Including Patients in Clinical Trials of the German Chronic Lymphocytic Leukemia Study Group (GCLLSG) or in "Real-Life" Outside of Clinical Trials. Anticancer Res. 2019 May;39(5):2591-2598. doi: 10.21873/anticanres.13382. PMID 31092457
- [Result] Eichhorst BF, Busch R, Obwandner T, Kuhn-Hallek I, Herschbach P, Hallek M; German CLL Study Group. Health-related quality of life in younger patients with chronic lymphocytic leukemia treated with fludarabine plus cyclophosphamide or fludarabine alone for first-line therapy: a study by the German CLL Study Group. J Clin Oncol. 2007 May 1;25(13):1722-31. doi: 10.1200/JCO.2006.05.6929. Epub 2007 Mar 26. PMID 17389338
- [Result] Eichhorst BF, Busch R, Hopfinger G, Pasold R, Hensel M, Steinbrecher C, Siehl S, Jager U, Bergmann M, Stilgenbauer S, Schweighofer C, Wendtner CM, Dohner H, Brittinger G, Emmerich B, Hallek M; German CLL Study Group. Fludarabine plus cyclophosphamide versus fludarabine alone in first-line therapy of younger patients with chronic lymphocytic leukemia. Blood. 2006 Feb 1;107(3):885-91. doi: 10.1182/blood-2005-06-2395. Epub 2005 Oct 11. PMID 16219797